CLINICAL TRIAL: NCT04282278
Title: Study of Anti-PD-1 Antibody Multimodal Combination as First-line Treatment on Time Window of Advanced Solid Tumor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Principal Investigator, Jian SHI, Principal Investigator, Hebei Medical University Fourth Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRHB-C001
Record Dates: First submitted 2020-02-18; First posted 2020-02-24 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental)
  Interventions: Drug: Camrelizumab/sintilimab+ Standard chemotherapy
- Group B (Experimental)
  Interventions: Drug: Camrelizumab/sintilimab+ apatinib（Intolerance to chemotherapy / refuse chemotherapy）
- Group C (Experimental)
  Interventions: Drug: Camrelizumab/sintilimab+ apatinib+ Standard chemotherapy

INTERVENTIONS:
Drug: Camrelizumab/sintilimab+ Standard chemotherapy — Camrelizumab/sintilimab：200mg，iv，30min，d4，q3w，24 months Standard chemotherapy：Researcher chooses standard treatment by recommended guidelines，d 1-3
  Arms: Group A
Drug: Camrelizumab/sintilimab+ apatinib（Intolerance to chemotherapy / refuse chemotherapy） — Camrelizumab/sintilimab：200mg，iv，30min，d4，q3w，24 months Apatinib：250mg，d1，qd，po
  Arms: Group B
Drug: Camrelizumab/sintilimab+ apatinib+ Standard chemotherapy — Camrelizumab/sintilimab：200mg，iv，30min，d7，q3w，24 months Apatinib：250mg，d1，qd，po Standard chemotherapy：Researcher chooses standard treatment by recommended guidelines，d 1-3
  Arms: Group C

SUMMARY:
The purpose of this study is to assess time window, efficacy and safety of patients who receive anti-PD-1 antibody multimodal combination as first-line treatment of advanced solid tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18 to 70 years old;
2. Patients with advanced solid tumors confirmed by histopathology or cytology and genetic testing was negative;
3. None previous chemotherapy, Antiangiogenic targeted therapy, Immune checkpoint inhibitors therapy（NOTE: neoadjuvant and adjuvant therapy is allowed）;
4. At least one measurable lesion (measuring≥10mm on spiral CT scan, satisfying the criteria in RECIST1.1);
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
6. Life expectancy greater than or equal to 18 weeks;
7. Major organ function has to meet the following certeria:

1) For results of blood routine test HB≥90g/L; ANC≥1.5×109/L; PLT≥90×109/L; 2) For results of blood biochemical test ALB≥30g/L ALT and AST<2.5×ULN, but<5×ULN if the transferanse elevation is due to liver metastases； TBIL≤1.5×ULN； Serum creatinine ≤1.5×ULN; 8. Left ventricular ejection fraction (LVEF) ≥50%; 9. Women of childbearing age must have contraceptive measures or have test pregnancy (serum or urine) enroll the study before 14 days, and the results must be negative, and take the methods of contraception during the test and the last to have drugs after 8 weeks. Men must be contraception or has sterilization surgery during the test and the last to have drugs after 8 weeks; 10. Participants were willing to join in this study, and written informed consent, good adherence, cooperate with the follow-up.

Exclusion Criteria:

1. Patients with symptomatic brain metastases;
2. Subjects with immunosuppressive medications within 14 days of first administration of study treatment, prednisone is used for less than 1 week, excluding nasal spray and inhaled corticosteroids or physiological doses of systemic steroid hormones (no more than 10 mg / day of prednisolone or other corticosteroids of equivalent pharmaceutical physiological dose);
3. The patient has any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, Hyperthyroidism; patients with vitiligo; Asthma has been completely relieved in childhood, and patients who do not need any intervention after adulthood can be included; asthma patients who require bronchodilators for medical intervention cannot be included);
4. Patients with other malignant tumors within 5 years (except for the treated skin basal cell carcinoma and cervical carcinoma in situ, dual or multiple primary tumors);
5. Human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS), active hepatitis B (HBV-DNA ≥1000 IU/ml) or hepatitis C (positive hepatitis C antibody, and HCV-RNA is higher than the lower limit of detection of the analytical method) or co-infection with hepatitis B and C, requiring antiviral treatment during the study ;
6. 3 months before study drug administration, the following occurred: myocardial infarction, severe / unstable angina pectoris, grade III-IV cardiac insufficiency according to New York Heart Association(NYHA) criteria, uncontrolled arrhythmias (including QTcF interval male> 450 ms, female> 470 ms ,The QTcF interval is calculated using Fridericia formula), symptomatic congestive heart failure, cerebrovascular accidents (including transient ischemic attack or symptomatic pulmonary embolism), in stable phase, need a cardiovascular physician evaluation;
7. Severe infections within 2 weeks before study drug administration (eg. Need intravenous drip antibiotics, antifungals or antivirals) or >38.5℃during screening visits or on the first scheduled day of dosing;
8. History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
9. Less than 4 weeks from the last clinical trial;
10. History of psychiatric drugs abuse and can't quit or patients with mental disorders;
11. The researchers think inappropriate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-07-16 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
PFS | evaluated in 24 months since the treatment began
  Baseline to measured date of progression or death from any cause

SECONDARY OUTCOMES:
ORR | tumor assessment every 6 weeks since the treatment began，up to 24 months
  Baseline to measured stable disease
DCR | tumor assessment every 6 weeks since the treatment began，up to 24 months
  Baseline to measured progressive disease
OS | the first day of treatment to death or last survival confirm date,up to 24 months
  Overall survival
Adverse events | up to 24 weeks
  Toxicity according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03. The number of Participants with adverse events will be recorded at each treatment visit.

CONTACTS AND LOCATIONS:
Overall Officials: Baoen Shan, Ph.D, Principal Investigator — Hebei Medical University Fourth Hospital; Jian Shi, Ph.D, Principal Investigator — Hebei Medical University Fourth Hospital
Locations (1):
- The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China